CLINICAL TRIAL: NCT07161635
Title: Post Market Clinical Evaluation of Clareon PanOptix Pro and Clareon PanOptix Pro Toric IOLs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILQ137-P001
Record Dates: First submitted 2025-09-02; First posted 2025-09-08 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Aphakia; Presbyopia
Keywords: Cataract; Eye Surgery
MeSH Terms: conditions — Aphakia; Presbyopia; Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Clareon PanOptix Pro/Pro Toric Trifocal IOL (Experimental): The clouded lens will be removed by phacoemulsification, after which the PanOptix Pro and/or PanOptix Pro Toric IOLs will be implanted.
  Interventions: Device: Clareon PanOptix Pro/Pro Toric Trifocal IOL; Procedure: Phacoemulsification

INTERVENTIONS:
Device: Clareon PanOptix Pro/Pro Toric Trifocal IOL — Intraocular lens (IOL) placed into the lens capsule of the eye during cataract surgery. IOLs are implantable medical devices intended for long-term use over the lifetime of the pseudophakic subject.
  Other Names: Clareon PanOptix Pro Trifocal IOL Models PXYWT0, PXCWT0, PXYAT0, PXCAT0; Clareon PanOptix Pro Trifocal Toric IOL Models PXYWT3- PXYWT6, PXCWT3-T6, PXYAT3-PXYAT6, PXCAT3-PXCAT6
Procedure: Phacoemulsification — Cataract surgery technique that uses ultrasound to break up and remove the clouded lens, allowing for IOL implantation.

SUMMARY:
The purpose of this study is to collect safety and performance data on two approved intraocular lenses (IOLs). This study will be conducted in participants who require cataract surgery in both eyes. The IOLs are designed to provide vision at far, arm's length, and near.

DETAILED DESCRIPTION:
Subjects will attend 9 scheduled study visits for a total individual duration of participation of approximately 7 months. Both eyes will undergo cataract surgery. The second eye surgery will occur within 7 to 14 days of the first.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects with cataracts in both eyes, planned for removal by routine surgery (phacoemulsification);
* Subject must be able to understand and sign an approved informed consent form;
* Subject is willing to complete all the required study visits for the duration of the study;
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Ocular conditions as specified in the protocol;
* Subjects who desire monovision correction;
* Previous intraocular or corneal surgery;
* Other protocol-defined exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Mean Binocular Photopic Best Corrected Distance Visual Acuity (BCDVA) | Month 1 and Month 6 postoperative
  Visual Acuity (VA) will be assessed for both eyes together (binocular) using Early Treatment Diabetic Retinopathy Study (ETDRS) reading charts at a distance of 4 meters from the subject under photopic (well-lit) conditions with correction in place. BCDVA will be measured in logarithm Minimum Angle of Resolution (logMAR). LogMAR values typically range from -0.3 (20/10 vision on the Snellen chart) to 1 (20/200 vision), with lower scores indicating better vision.

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Principal Clinical Trial Operations, Surgical, Study Director — Alcon Research LLC
Locations (5):
- United States (5):
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Moyes Eye Center, Kansas City, Missouri
  - Carolina Eyecare Physicians LLC, Mt. Pleasant, South Carolina
  - Houston Eye Associates, Houston, Texas
  - The Eye Institute of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No